CLINICAL TRIAL: NCT02462213
Title: The Influence of Amyloid Protein on Myocardial Tissue Characteristics and Function: Prognostic and Diagnostic Significance of Cardiac Magnetic Resonance Findings
Brief Title: Prospective Identification of Cardiac Amyloidosis by Cardiac Magnetic Resonance Imaging
Acronym: PICA-CMR
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit patients who had not had MRI first.
Sponsor: University of Cincinnati (Other)
Collaborators: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Robert O'Donnell, Associate Professor, University of Cincinnati
Other Study IDs: 2013-3043
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Amyloidosis; Paraproteinemias; Cardiomyopathies
Keywords: Cardiac amyloidosis; Cardiac MRI; Infiltrative cardiomyopathies
MeSH Terms: conditions — Amyloidosis; Paraproteinemias; Cardiomyopathies; Amyloid Neuropathies, Familial | interventions — Amyloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Amyloidosis: Patients being managed for amyloidosis without prior history of cardiac involvement
  Interventions: Other: Amyloidosis
- Cardiac amyloidosis: Patients being managed for cardiac amyloidosis
  Interventions: Other: Cardiac Amyloidosis

INTERVENTIONS:
Other: Amyloidosis — Patients with amyloidosis without cardiac involvement will undergo cardiac MRI and possible biochemical analysis during the course of the study.
  Groups: Amyloidosis
Other: Cardiac Amyloidosis — Patients with confirmed cardiac amyloidosis will undergo cardiac MRI and possible biochemical analysis during the course of the study.
  Groups: Cardiac amyloidosis

SUMMARY:
Cardiac amyloidosis describes a process by which abnormally folded proteins infiltrate the heart tissue. Given the insidious nature of this disease process, diagnosis is often too late for a meaningful intervention. Advances in the treatment of the amyloidoses have improved outcomes for patients with these conditions. The focus of this study is to identify the involvement of the heart, most closely associated with mortality, so that aggressive management can be instituted improving prognosis.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL

Hypothesis:

The presence of amyloid protein in the myocardium changes its function and tissue characteristics. These changes are responsible for the poor prognosis of patients with cardiac amyloidosis. Cardiac magnetic resonance imaging (CMR) offers a novel, non-invasive approach to identify cardiac involvement that may impact patient management. This study will include the prospective validation of CMR parameters qualified as being abnormal in the retrospective study (study ID 2012-3315) and the current literature. The myocardium/blood pool inversion time null point ratio (Myo/BlP TI0 ratio), has been qualified as being significantly different when compared to controls in the retrospective study.

Specific Aims:

1. Validate the diagnostic accuracy of CMR parameters in a prospective manner for cardiac amyloidosis patients.
2. CMR parameters, including the Myo/BlP TI0 ratio, will be compared to serum biomarkers (TroponinT, NT-proBNP, serum lambda/kappa free light chain concentration), established to have prognostic value in cardiac amyloidosis. Subjects will be followed via death registry and/or medical records to compare the prognostic value of the CMR parameter with the biomarkers.
3. CMR parameters will be used to assess for the presence of early cardiac involvement in amyloidosis patients without clinically apparent cardiac involvement (as determined by symptoms, biomarkers and/or cardiac imaging).
4. CMR will be used to follow patients undergoing treatment, when available, to determine whether CMR parameters consistent with the presence of cardiac amyloidosis, change during treatment.

Background and Significance:

Matthias Schleiden, a German botanist and co-creator of the cell theory, used the term amyloid in 1834 to characterize the waxy starch in plants. Today, amyloid is used to describe any of a number of small proteins which when aggregated lead to insoluble fibrillar deposits. Many mechanisms of protein dysfunction contribute to amyloidogenesis, including "non-physiologic proteolysis, defective physiologic proteolysis, mutations involving changes in thermodynamic or kinetic properties, and pathways that are yet to be defined". Amyloid deposits are identified on the basis of their apple-green birefringence under a polarized light microscope after staining with Congo red. They can also be identified based on the presence of rigid, non-branching fibrils using electron microscopy. Amyloidosis describes the infiltration of organs by these insoluble deposits. In humans, about 27 different unrelated proteins are known to form amyloid fibrils in vivo. The organs involved and clinical presentations are dependent on the precursor protein. A small number of the amyloidoses can have cardiac involvement with a significant impact on mortality. The clinically most significant cardiac amyloidoses include immunoglobulin light chain amyloidosis (AL) and the transthyretin amyloidoses (ATTR); ATTR being either hereditary secondary to mutations in the transthyretin gene or acquired secondary to wild type transthyretin protein.

AL amyloidosis, the most common type of systemic amyloidosis, is associated with plasma cell dyscrasias. In AL amyloidosis, fifty percent of affected patients will have cardiac involvement. Despite the potential for amyloid deposition in multiple organs, cardiac involvement continues to dictate the poorest prognosis. Once congestive heart failure develops in a patient with AL amyloidosis, survival is less than 6 months if untreated. Therefore, patients with AL amyloidosis are screened, by assessing serum troponins and brain natriuretic peptides, to determine whether cardiac involvement is present. Patients with ATTR amyloidosis typically has a more insidious onset in comparison. ATTR amyloidosis also responds better to traditional congestive heart failure management. However, neither AL nor the ATTR amyloidoses are managed like traditional heart failure making appropriate diagnosis critical for best care. Furthermore, early diagnosis of cardiac involvement may improve outcomes but requires heightened suspicion and a systematic clinical approach to evaluation [3].

In cardiac amyloidosis, there can be evidence of disease on routine testing. Restrictive physiology by echocardiography, low EKG voltage as well as additional EKG abnormalities are often identified in advanced cardiac amyloidosis. Routine nuclear cardiac imaging has not proven to be helpful in diagnosis, although 123I-MIBG does appear to demonstrate co-localization of denervation with amyloid deposition. Unfortunately, no routine cardiac testing is specific for cardiac amyloidosis. Therefore, in the absence of high clinical suspicion for cardiac amyloidosis, the appropriate diagnosis will often be missed.

Endomyocardial biopsy remains the gold standard for making the diagnosis of cardiac involvement. However, given the invasive nature of endomyocardial biopsy and associated risks (including death), the diagnosis of cardiac amyloidosis is usually made by non-invasive means; this diagnosis being supported by a non-cardiac biopsy demonstrating amyloid deposits. The most frequently biopsied site is the abdominal fat pad, usually positive in patients with AL amyloidosis. However, ATTR amyloidosis is not reliably identified with fat pad biopsy. Therefore, a negative fat pad biopsy requires further work up including endomyocardial biopsy with associated immunostaining and genetic testing for transthyretin mutations. Supporting the diagnosis of cardiac amyloidosis by noninvasive techniques such as EKG, echocardiography and serum amyloid component scintigraphy has been shown to have significant limitations. A novel non-invasive approach is required to ensure accurate diagnosis. Given the limitations of previously used non-invasive techniques, there has been interest over the last decade in using cardiovascular magnetic resonance (CMR) imaging in the diagnosis of cardiac amyloidosis.

The utility of CMR in evaluating patients with cardiac amyloidosis was first proposed in the 1990s. However, evaluation was limited to the assessment of myocardial morphology and function. It was not until the turn of the century that the powerful diagnostic potential of delayed gadolinium enhancement (DGE) was realized. The first utility of DGE was in the evaluation of myocardial viability in patients with coronary artery disease. It quickly became apparent that DGE could also be used to evaluate patients with non-ischemic cardiomyopathies. The characterization of cardiac amyloidosis with DGE was first described as global sub-endocardial enhancement. Abnormal T1 transmyocardial maps were used to both describe the abnormality and to assist in the determination of prognosis. However, these studies were limited by inclusion of only patients with biopsy-proven amyloidosis who also met the echocardiographic criteria for restrictive physiology, common to advanced cardiac amyloidosis. More recent work precluding the use of echocardiographic diagnosis supported the concept that the inability to null the myocardium relative to the blood pool may be an early sign of cardiac amyloidosis. In addition, to the DGE data, studies have utilized T1 and T2 weighted imaging to identify abnormal extracellular volume (ECV) and myocardial edema in the cardiac amyloidosis population.

It has been the culmination of these findings, in addition to our own experience studying cardiac amyloidosis that led to the hypothesis that the presence of amyloid protein, known to increase the ECV, may also change the inversion time curves of both the blood pool and the myocardium. These features, as well as abnormal functional parameters, will help detect cardiac amyloidosis earlier than would otherwise be possible by morphologic assessment. The possibility of diagnosing sub-clinical disease has implications for screening patients with known amyloidosis for early cardiac involvement. Also, CMR parameters may be useful in assessing response to treatment of the plasma cell dyscrasias, such as cardiac amyloidosis, that may be complicated by heart failure and ventricular tachycardia. Lastly, the relationship of the MRI findings to cardiac biomarkers has yet to be described and will be assessed in this study.

Preliminary Data:

The investigators have observed a significant difference between the Myo/BlP TI0 ratio in patients with cardiac amyloidosis when compared with controls both with preserved LV function (CTL) and non-amyloid cardiomyopathies (CTL-CMP). The Myo/BlP TI0 ratio of the CA group is close to 1 to 1 (0.95 +/- 0.16) leading to poor myocardium and blood pool contrast in the corresponding delayed enhancement images acquired following the TI scout (Figure 7). The Myo/BlP TI0 ratio provides a quantitative method to support the diagnosis of cardiac amyloidosis in patients presenting with cardiac symptoms.

Estimated Period of Time to Completion:

Estimated time to completion of aim 1, 2 and 4 will depend on power calculations following the acquisition of pilot prospective data. The estimated timing of completion of aim 3 will be 12-18 months from the start of data acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting diagnostic criteria for the target population will be recruited for the study. Age range will be 18 to 85 years of age.

Exclusion Criteria:

* Exclusion criteria will include history of heart transplantation as well as any contraindications for 1.5T CMR. For the use of GBCA, patients with acute renal failure or stage IV/V chronic renal failure will be excluded. Patients with end stage renal failure receiving peritoneal dialysis will also be excluded. Women who are pregnant or breast feeding will also be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with amyloidosis will be recruited from the hematology clinic from participating institutions. Patients with confirmed cardiac amyloidosis will be recruited from either the cardiology or hematology clinics of participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identification of cardiac amyloidosis using contrast cardiovascular MRI | 2 years

SECONDARY OUTCOMES:
All cause mortality | two years

CONTACTS AND LOCATIONS:
Overall Officials: Robert E O'Donnell, MD MSc, Principal Investigator — University of Cincinnati; Jennifer Daniels, MSc, Study Director — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Buxbaum JN. The systemic amyloidoses. Curr Opin Rheumatol. 2004 Jan;16(1):67-75. doi: 10.1097/00002281-200401000-00013. PMID 14673392
- [Background] Merlini G, Bellotti V. Molecular mechanisms of amyloidosis. N Engl J Med. 2003 Aug 7;349(6):583-96. doi: 10.1056/NEJMra023144. No abstract available. PMID 12904524
- [Background] Shah KB, Inoue Y, Mehra MR. Amyloidosis and the heart: a comprehensive review. Arch Intern Med. 2006 Sep 25;166(17):1805-13. doi: 10.1001/archinte.166.17.1805. PMID 17000935
- [Background] Falk RH. Diagnosis and management of the cardiac amyloidoses. Circulation. 2005 Sep 27;112(13):2047-60. doi: 10.1161/CIRCULATIONAHA.104.489187. No abstract available. PMID 16186440
- [Background] Dubrey SW, Cha K, Anderson J, Chamarthi B, Reisinger J, Skinner M, Falk RH. The clinical features of immunoglobulin light-chain (AL) amyloidosis with heart involvement. QJM. 1998 Feb;91(2):141-57. doi: 10.1093/qjmed/91.2.141. PMID 9578896
- [Background] Kyle RA, Gertz MA. Primary systemic amyloidosis: clinical and laboratory features in 474 cases. Semin Hematol. 1995 Jan;32(1):45-59. No abstract available. PMID 7878478
- [Background] Klein AL, Cohen GI. Doppler echocardiographic assessment of constrictive pericarditis, cardiac amyloidosis, and cardiac tamponade. Cleve Clin J Med. 1992 May-Jun;59(3):278-90. doi: 10.3949/ccjm.59.3.278. PMID 1516216
- [Background] Noordzij W, Glaudemans AW, van Rheenen RW, Hazenberg BP, Tio RA, Dierckx RA, Slart RH. (123)I-Labelled metaiodobenzylguanidine for the evaluation of cardiac sympathetic denervation in early stage amyloidosis. Eur J Nucl Med Mol Imaging. 2012 Oct;39(10):1609-17. doi: 10.1007/s00259-012-2187-8. Epub 2012 Jul 18. PMID 22806059
- [Background] Maceira AM, Joshi J, Prasad SK, Moon JC, Perugini E, Harding I, Sheppard MN, Poole-Wilson PA, Hawkins PN, Pennell DJ. Cardiovascular magnetic resonance in cardiac amyloidosis. Circulation. 2005 Jan 18;111(2):186-93. doi: 10.1161/01.CIR.0000152819.97857.9D. Epub 2005 Jan 3. PMID 15630027
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] McCrohon JA, Moon JC, Prasad SK, McKenna WJ, Lorenz CH, Coats AJ, Pennell DJ. Differentiation of heart failure related to dilated cardiomyopathy and coronary artery disease using gadolinium-enhanced cardiovascular magnetic resonance. Circulation. 2003 Jul 8;108(1):54-9. doi: 10.1161/01.CIR.0000078641.19365.4C. Epub 2003 Jun 23. PMID 12821550
- [Background] vanden Driesen RI, Slaughter RE, Strugnell WE. MR findings in cardiac amyloidosis. AJR Am J Roentgenol. 2006 Jun;186(6):1682-5. doi: 10.2214/AJR.04.0871. PMID 16714659
- [Background] Maceira AM, Prasad SK, Hawkins PN, Roughton M, Pennell DJ. Cardiovascular magnetic resonance and prognosis in cardiac amyloidosis. J Cardiovasc Magn Reson. 2008 Nov 25;10(1):54. doi: 10.1186/1532-429X-10-54. PMID 19032744
- [Background] Syed IS, Glockner JF, Feng D, Araoz PA, Martinez MW, Edwards WD, Gertz MA, Dispenzieri A, Oh JK, Bellavia D, Tajik AJ, Grogan M. Role of cardiac magnetic resonance imaging in the detection of cardiac amyloidosis. JACC Cardiovasc Imaging. 2010 Feb;3(2):155-64. doi: 10.1016/j.jcmg.2009.09.023. PMID 20159642
- [Background] Krombach GA, Hahn C, Tomars M, Buecker A, Grawe A, Gunther RW, Kuhl HP. Cardiac amyloidosis: MR imaging findings and T1 quantification, comparison with control subjects. J Magn Reson Imaging. 2007 Jun;25(6):1283-7. doi: 10.1002/jmri.20917. PMID 17520735
- [Background] Guglin M, Aljayeh M, Saiyad S, Ali R, Curtis AB. Introducing a new entity: chemotherapy-induced arrhythmia. Europace. 2009 Dec;11(12):1579-86. doi: 10.1093/europace/eup300. Epub 2009 Oct 3. PMID 19801562
- [Background] Shakir DK, Rasul KI. Chemotherapy induced cardiomyopathy: pathogenesis, monitoring and management. J Clin Med Res. 2009 Apr;1(1):8-12. doi: 10.4021/jocmr2009.02.1225. Epub 2009 Mar 24. PMID 22505958
- [Background] Dispenzieri A, Lacy MQ, Katzmann JA, Rajkumar SV, Abraham RS, Hayman SR, Kumar SK, Clark R, Kyle RA, Litzow MR, Inwards DJ, Ansell SM, Micallef IM, Porrata LF, Elliott MA, Johnston PB, Greipp PR, Witzig TE, Zeldenrust SR, Russell SJ, Gastineau D, Gertz MA. Absolute values of immunoglobulin free light chains are prognostic in patients with primary systemic amyloidosis undergoing peripheral blood stem cell transplantation. Blood. 2006 Apr 15;107(8):3378-83. doi: 10.1182/blood-2005-07-2922. Epub 2006 Jan 5. PMID 16397135